CLINICAL TRIAL: NCT03825315
Title: A Phase II, Prospective, Randomized, Double-Blind, Multi-center, Placebo-Controlled Trial of DaxibotulinumtoxinA for Injection for the Management of Plantar Fasciitis
Brief Title: DaxibotulinumtoxinA for Injection for the Treatment of Plantar Fasciitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1820201
Record Dates: First submitted 2019-01-15; First posted 2019-01-31 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Plantar Fasciitis
Keywords: DAXI for injection,; Plantar Fasciitis,; Heel Pain,; BotulinumtoxinA
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to 1 of 3 treatment groups: DAXI for injection LOW dose, DAXI for injection HIGH dose, Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DAXI 80 U (Experimental): LOW Dose Group
  Interventions: Biological: DAXI 80 U
- DAXI 120 U (Experimental): HIGH Dose Group
  Interventions: Biological: DAXI 120 U
- Placebo (Placebo Comparator): Placebo Group.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: DAXI 80 U — DaxibotulinumtoxinA for injection for the treatment of unilateral plantar fasciitis (PF) with 80 U (Low Dose Group)
  Arms: DAXI 80 U
Biological: DAXI 120 U — DaxibotulinumtoxinA for injection for the treatment of unilateral plantar fasciitis (PF) 120 U (High Dose Group)
  Arms: DAXI 120 U
Other: Placebo — Placebo is a sterile lyophilized product consisting of inactive ingredients without the neurotoxin to be reconstituted with sterile, non-preserved 0.9% sodium chloride solution.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel group, multi-center trial of a single administration of DaxibotulinumtoxinA (DAXI) (high-dose; low-dose) for injection versus placebo for the management of Plantar Fasciitis.

DETAILED DESCRIPTION:
Approximately 150 subjects, recruited from approximately 20 study centers in the United States (US) will be randomized to DAXI (HIGH-dose; LOW-dose) or placebo group, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, including authorization to release health information.
* Male or female subjects 18 to 65 years of age with diagnosis of unilateral plantar fasciitis.
* Persistent heel pain.
* Women of child bearing potential must have a negative pregnancy test at Screening and Injection Visits and must use an effective method of contraception during the course of the study.

Exclusion Criteria:

* Previous injection of botulinum toxin in the lower extremities or feet.
* Previously suffered a partial or full thickness tear or surgery of the plantar fascia within the 5 years preceding participation in the investigation.
* Pregnant, nursing, or planning a pregnancy during the study.
* Current enrollment in an investigational drug or device study or participation in such a study within the last 30 days prior to first visit.
* Any condition or situation which, in the Investigator's opinion, puts the subject at significant risk, could confound the trial results, or may interfere significantly with the subject's participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Aung Foot Health Clinic, Tucson, Arizona
  - Sacramento Foot and Ankle Center, Inc, Carmichael, California
  - Bay Area Foot Care, Castro Valley, California
  - West Coast Foot and Ankle, Huntington Beach, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Bay Area Foot Care, San Francisco, California
  - University Foot and Ankle Foundation, Santa Monica, California
  - LA Podiatry Group, West Palm Beach, Florida
  - Podiatry 1st, Belleville, Illinois
  - Rosalind Franklin University of Medicine & Science, North Chicago, Illinois
  - Kansas Institute of Research, Overland Park, Kansas
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - Medical Research International, Oklahoma City, Oklahoma
  - North Texas Institute of Neurology and Headache, Frisco, Texas
  - Hermann Drive Research Hospital, Houston, Texas
  - Futuro Clinical Trials, LLC, McAllen, Texas
  - Strash Foot and Ankle Care, San Antonio, Texas
  - The Podiatry Group of South Texas, San Antonio, Texas
  - Rocky Mountain Foot and Ankle, LLC, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DAXI 80 U | DAXI 120 U | Placebo
Started | 49 | 54 | 52
Completed | 42 | 48 | 46
Not Completed | 7 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- DAXI 120 U: DaxibotulinumtoxinA for injection for the treatment of unilateral plantar fasciitis (PF) with 120 U (High Dose Group)
- Total: Total of all reporting groups
Arm/Group | DAXI 80 U | DAXI 120 U | Placebo | Total
Number analyzed (Participants) | 49 | 54 | 52 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (9.06) | 47.1 (8.17) | 48.5 (8.02) | 48.1 (8.38)
Age, Customized [Count of Participants; unit: Participants]
  <= 50 years | 26 | 34 | 34 | 94
  > 50 years | 23 | 20 | 18 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 36 | 103
  Male | 14 | 22 | 16 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Black | 3 | 4 | 3 | 10
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  White | 44 | 44 | 47 | 135
  Multiple | 0 | 0 | 0 | 0
  Other | 0 | 1 | 0 | 1
  Not reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 8 in the Numeric Pain Rating Scale (NPRS) Score
Description: Change from baseline in the Numeric Pain Rating Scale (NPRS) score, which is recorded within 15 minutes after stepping out of bed in the morning and averaged over 5 days (defined as 4 days prior to study visit and on the study visit day), at Week 8.
  The outcome was measured by an 11-point scale scored from 0-10 where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: Week 8
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DAXI 80 U | DAXI 120 U | Placebo
Number analyzed (Participants) | 49 | 54 | 52
score on a scale | -3.29 (0.329) | -3.25 (0.298) | -2.75 (0.302)

2. Secondary Outcome: Change From Baseline at Week 8 in Foot Function Index (FFI)
Description: The Foot Function Index (FFI) is a 23 item questionnaire divided into 3 subscales measuring pain, disability, and activity restriction. The scale was scored from 0 (no pain) to 10 (worst pain imaginable). Both total and sub-scale scores are produced.
  The total FFI equals the average of the 3 subscale scores. Pain, disability, and activity limitation subscale scores were normalized and the range is from 0 to 100. The total FFI equals the average of the 3 subscale scores. Pain, disability, and activity limitation subscale scores range from 0 to 100.
Time Frame: Week 8
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | DAXI 80 U | DAXI 120 U | Placebo
Number analyzed (Participants) | 49 | 54 | 52
score on a scale | -29.02 (2.202) | -27.37 (2.149) | -23.63 (2.185)

3. Secondary Outcome: Proportion of Subjects With a Decrease From Baseline of >= 20% in NPRS
Description: For the proportion of subjects with a decrease from baseline of >= 20% in NPRS score at Week 8
Time Frame: Week 8
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | DAXI 80 U | DAXI 120 U | Placebo
Number analyzed (Participants) | 49 | 54 | 52
Participants | 35 | 41 | 34

ADVERSE EVENTS:
Time Frame: The adverse events were collected throughout the entire study, through week 24.
Description: The Safety Population includes all subjects who received at least 1 study treatment injection and was used to assess AEs and SAEs
Arm/Group | DAXI 80 U | DAXI 120 U | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/54 | 0/52
Serious Adverse Events (participants affected / at risk) | 2/49 | 2/54 | 0/52
Other Adverse Events (participants affected / at risk) | 7/49 | 12/54 | 10/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAXI 80 U (N=49) | DAXI 120 U (N=54) | Placebo (N=52)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAXI 80 U (N=49) | DAXI 120 U (N=54) | Placebo (N=52)
Nasopharyngitis (Infections and infestations) | 2 (3) | 3 (3) | 3 (5)
Influenza (Infections and infestations) | 2 (2) | 4 (4) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Injection site pain (General disorders) | 3 (3) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study Center and/or Investigator shall submit to Revance a copy of the proposed publication at least sixty (60) days prior to the submission thereof for publication or disclosure to a third party: (i)to provide Revance with the opportunity to review and comment on the contents thereof, (ii)to identify any Confidential Information to be deleted from the proposed publication or disclosure, and (iii)or delay the publication or disclosure 90 days to allow Revance to pursue patent protections.

DOCUMENTS (2):
  • Study Protocol (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03825315/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT03825315/SAP_001.pdf